CLINICAL TRIAL: NCT04654351
Title: A Multicenter, Open-Label, Non-randomized Phase 3 Study to Assess the Safety, Efficacy and Pharmacokinetics of Subcutaneous Administration of Icatibant (TAK-667) in Japanese Children and Adolescents With Acute Attacks of Hereditary Angioedema
Brief Title: A Study of Icatibant (TAK-667) in Japanese Children and Teenagers With Acute Attacks of Hereditary Angioedema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-667-3001; U1111-1260-2627 (Other: WHO); jRCT2041200073 (Registry Identifier: jRCT)
Record Dates: First submitted 2020-11-29; First posted 2020-12-04 (Actual); Results first posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-01

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — icatibant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAK-667 (Experimental): TAK-667, single SC administration on the abdomen on Day 1. The dose of TAK-667 will be dependent on the participant's body weight (Up to 30 mg; 10 mg for 12 kg to 25 kg, 15 mg for 26 kg to 40 kg, 20 mg for 41 kg to 50kg, 25 mg for 51 kg to 65 kg, 30 mg for >65 kg).
  Interventions: Drug: TAK-667

INTERVENTIONS:
Drug: TAK-667 — TAK-667 single SC administration
  Other Names: Icatibant

SUMMARY:
The main aim of the study is to check for side effects from icatibant in children and teenagers with hereditary angioedema (HAE). Other aims are to check how well icatibant controls HAE symptoms in these children and teenagers, and how much icatibant stays in their blood.

At the first visit, the study doctor will check if each child or teenager can take part. For those who can take part, participants and their parents or caregivers will visit the clinic or hospital when they have their next HAE attack. Participants will receive 1 injection (shot) of icatibant in a vein and will stay at the clinic or hospital until their HAE symptoms are under control. Participants can receive up to 2 more injections of icatibant over time if their HAE symptoms don't improve or get worse.

After the participants go home, the study staff will follow up with them by a telephone call 1 to 2 days later. Then, the participants will visit the clinic or hospital 1 week after they received the icatabant injection.

The participant can visit the clinic or hospital and be treated with icatibant in the same way for up to 3 HAE attacks in total.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-667. TAK-667 is being tested to treat Japanese Children and Adolescents who experience acute attack of HAE. This study will look at safety, efficacy and pharmacokinetics (PK) of people who take TAK-667.

The study will enroll at least up to 3 participants. Participants will take TAK-667 with SC administration on the abdomen. The dose of TAK-667 will be dependent on the participant's body weight (Up to 30 mg; 10 mg for 12 kg to 25 kg, 15 mg for 26 kg to 40 kg, 20 mg for 41 kg to 50kg, 25 mg for 51 kg to 65 kg, 30 mg for >65 kg).

This multi-center trial will be conducted in Japan. The overall time to participate in this study is 25 days as a maximum (screening day for initial attack plus 8 days post dose for each 3 attacks as a maximum). Participants will make multiple visits to the clinic and will be closely monitored in the hospital/study center for at least 8 hours after administration and receive physical examination and assessment to evaluate safety, efficacy and PK. Hospitalization may be prolonged until, in the opinion of the investigator, the participant is clinically stable and onset of HAE attack is completely resolved.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator or subinvestigator, the participant's parent or legal guardian is capable of understanding and complying with protocol requirements.
2. The participant's parent or the participant's legal guardian is capable of signing and dating a written informed consent form on behalf of the participant prior to the initiation of any study procedures. Written informed assent is also obtained from the participant as much as possible.
3. The participant is in Japan and is Japanese; defined as born in Japan and having Japanese parents and Japanese maternal and paternal grandparents.
4. The participant is male or female and 2 to <18 years of age (ie, from the second birthday through the day prior to the eighteenth birthday) at the time of informed consent.
5. The participant weighs >=12 kg at the time of the current HAE attack.
6. The participant who has a documented and confirmed diagnosis of HAE type I or II. Diagnosis may be based on historical data using the following criteria:

   1. Family history of angioedema
   2. Characteristic attack manifestations, recurrent attacks
   3. Functional complement 1 (C1) esterase inhibitor (C1-INH) deficiency
   4. In the absence of a family history of angioedema, exclusion of other forms of angioedema (eg. angiotensin converting enzyme (ACE)-induced angioedema, allergic angioedema) based on medical judgement (eg, concomitant medication, response to antihistamines or glucocorticoids, information of genetic mutation).
7. If the participant does not have a documented and confirmed diagnosis of HAE type I or II based on historical data, including C1-INH deficiency, the participant's diagnosis must be determined prior to treatment by C1-INH test results which demonstrate a functional C1-INH deficiency.

   1. HAE type I: Low amount of C1-INH protein and low level of C1-INH activity; HAE type II: Normal or increased amount of C1-INH protein and low level of C1-INH activity
   2. In the absence of a family history of angioedema, exclusion of other forms of angioedema (eg. ACE-induced angioedema, allergic angioedema) based on medical judgement (eg, concomitant medication, response to antihistamines or glucocorticoids, information of genetic mutation).
8. The current HAE attack must be in the cutaneous, abdominal, and/or laryngeal (inclusive of laryngeal and pharyngeal) areas, but no prespecified attack severity criteria are required for treatment.
9. The participant commences treatment within 12 hours after the onset of current HAE attack.
10. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study, and proves negative in the pregnancy test at screening.

Exclusion Criteria:

1. The participant will require an intervention to support the airway (eg, intubation, tracheotomy, cricothyrotomy) due to the current HAE attack.
2. The participant presents with an HAE attack with laryngeal/upper respiratory tract symptoms which are considered severe in the investigator's clinical judgment and which may necessitate urgent care and/or impede the conduct of study efficacy assessments.
3. The participant has a diagnosis of angioedema other than HAE
4. The participant has evidence of stroke or coronary artery disease based on medical history at the screening examination or at pretreatment; eg, acute ischemic heart disease, unstable angina pectoris, severe coronary heart disease or congestive heart failure, that in the investigator's judgment would be a contraindication for participation in the trial (New York Heart Association [NYHA] class 3 and 4).
5. The participant has received treatment with any pain medication since the onset of the current HAE attack.
6. The participant has received replacement therapy (C1-INH products, fresh frozen plasma [FFP]) within 5 days (120 hours) from the onset of the current HAE attack.
7. The participant has received treatment with ACE inhibitors within 7 days prior to treatment.
8. The participant has used hormonal contraceptive within 90 days prior to treatment.
9. The participant has received androgen or attenuated androgens (eg, danazol, testosterone) within 90 days prior to treatment.
10. The participant has participated in another clinical study within the past 30 days before screening.
11. The participant, the participant's parent, or legal guardian is unable to understand the nature, scope, and possible consequences of the protocol, or is unlikely to comply with the protocol assessments, unable to return for follow up visits, or unlikely to complete the study for any reason.
12. If female, the participant is pregnant or lactating or intending to become pregnant before participating in this study, during the study, and within 30 days after last dose of the icatibant.
13. The participant has a history of hypersensitivity or allergies to icatibant.
14. The participant is judged by the investigator as being ineligible for any other reason; eg. a serious concomitant illness or condition.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- Japan (3):
  - Aich Medical University Hospital, Nagakute, Aichi-ken
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Kagoshima University Hospital, Kagoshima

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5ff6d454565ce300294c6abc

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in Japan from 15 January 2021 to 27 July 2021.
Pre-assignment Details: Participants with a diagnosis of hereditary angioedema (HAE) type I or II were enrolled in a single arm to receive TAK-667 single-dose per attack. Up to two additional injections were permitted per attack. Participants who subsequently experienced an acute attack continued to receive TAK-667 for up to a total of three eligible icatibant-treated attacks.
Groups:
- TAK-667 10-30 mg: TAK-667 five-weight-band dosing of up to maximum of 10-30 mg injection, subcutaneously (SC), once on Day 1, and if necessary (there was insufficient relief or worsening of symptoms), up to two additional doses with a time interval of at least 6 hours between doses within 48 hours of initial injection per attack for up to 3 HAE attacks till the end of study (approximately 6 months). The dose of TAK-667 depended upon the participant's body weight (10 mg for 12 kg to 25 kg, 15 mg for 26 kg to 40 kg, 20 mg for 41 kg to 50kg, 25 mg for 51 kg to 65 kg, 30 mg for >65 kg).
Period: Overall Study
Arm/Group | TAK-667 10-30 mg
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- TAK-667 10-30 mg: TAK-667 five-weight-band dosing of up to maximum of 30 mg injection, SC, once on Day 1, and if necessary (there was insufficient relief or worsening of symptoms), up to two additional doses with a time interval of at least 6 hours between doses within 48 hours of initial injection per attack for up to 3 HAE attacks till the end of study (approximately 6 months). The dose of TAK-667 depended upon the participant's body weight (10 mg for 12 kg to 25 kg, 15 mg for 26 kg to 40 kg, 20 mg for 41 kg to 50kg, 25 mg for 51 kg to 65 kg, 30 mg for >65 kg).00
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Due to risk of identification, data for age is not reported to protect participant privacy.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Due to risk of identification, data for gender is not reported to protect participant privacy.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to risk of identification, data for ethnicity is not reported to protect participant privacy.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to risk of identification, data for race is not reported to protect participant privacy.
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced at Least One Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. A treatment-emergent adverse event (TEAE) was defined as any adverse event occurring after the start of Icatibant administration of the treatment period.
Time Frame: Up to approximately 6 months
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- TAK-667 10-30 mg: TAK-667 five-weight-band dosing of up to maximum of 30 mg injection, SC, once on Day 1, and if necessary (there was insufficient relief or worsening of symptoms), up to two additional doses with a time interval of at least 6 hours between doses within 48 hours of initial injection per attack for up to 3 HAE attacks till the end of study (approximately 6 months). The dose of TAK-667 depended upon the participant's body weight (10 mg for 12 kg to 25 kg, 15 mg for 26 kg to 40 kg, 20 mg for 41 kg to 50kg, 25 mg for 51 kg to 65 kg, 30 mg for >65 kg).
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
Participants | 0

2. Primary Outcome: Number of Participants With Injection Site Reactions
Description: Injection sites were examined for erythema, swelling, cutaneous pain, burning sensation, itching/pruritus, and warm sensation. Data for injection site reactions were collected separately from general reports of AEs. As pre-defined in the protocol, an injection site reaction not meeting SAE criteria was not required to be reported additionally as an AE.
Time Frame: Postdose, up to Day 8
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
percentage of participants | 2

3. Secondary Outcome: Number of Participants Who Experienced at Least One TEAE Related to Resting 12-lead Electrocardiogram
Description: An AE means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. A TEAE was defined as any AE occurring after the start of Icatibant administration of the Treatment Period. A resting 12-lead ECG was recorded and reported for participants shifts from within normal limits at baseline to abnormal, but not clinically significant, or abnormal and clinically significant after study drug administration.
Time Frame: Up to approximately 6 months
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
Participants | 0

4. Secondary Outcome: Number of Participants Who Experienced at Least One TEAE Related to Vital Sign
Description: An AE means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. A TEAE was defined as any AE occurring after the start of Icatibant administration of the Treatment Period. Vital signs included body temperature (oral), sitting blood pressure (after 5 minutes resting), respiration rate and pulse (beats per minute [bpm]).
Time Frame: Up to approximately 6 months
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
Participants | 0

5. Secondary Outcome: Number of Participants Who Experienced at Least One TEAE Related to Clinical Laboratory Parameters
Description: An AE means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. A TEAE was defined as any AE occurring after the start of Icatibant administration of the Treatment Period. The laboratory parameters included hematology, serum chemistries, and urinalysis.
Time Frame: Up to approximately 6 months
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
Participants | 0

6. Secondary Outcome: Number of Participants Who Experience at Least One TEAE Related to Clinically Significant Changes in Reproductive Hormones
Description: An AE means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. A TEAE was defined as any AE occurring after the start of Icatibant administration of the Treatment Period. Blood samples were collected to assess follicle stimulating hormone (FSH), luteinizing hormone (LH), estradiol, and progesterone in females, and FSH, LH, and testosterone in males.
Time Frame: Up to approximately 6 months
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
Participants | 0

7. Secondary Outcome: Number of Participants Who Reported Presence of Anti-icatibant Antibodies
Description: Serum samples for immunogenicity testing were collected for determination of anti-icatibant antibodies. If hypersensitivity was observed, it was reported as an AEs of special interest. An AE means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product.
Time Frame: Up to approximately 6 months
Population: Safety analysis set was defined as all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
Participants | 0

8. Secondary Outcome: Time to Onset of Symptom Relief With Investigator-Rated Symptom Scores Assessed by Investigator
Description: The time to onset of symptom relief, defined as the duration of time in hours from the time of icatibant administration to the earliest time at which at least a 20% improvement is observed in the average post-treatment score with no worsening of any single component score. Investigator-rated symptom score was used for assessment and scoring of cutaneous, abdominal, and laryngeal symptoms of acute HAE attacks related to daily activities. The score ranged from 0 to 4 and each number of scores meant the following: 0 = none; absence of symptoms, 1 = mild (no to mild interference with daily activities), 2 = moderate (moderate interference with daily activities), 3 = severe (severe interference with daily activities), 4 = very severe (very severe interference with daily activities).
Time Frame: Baseline, and post dose on Day 1
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: hours
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
hours | NA [0.9 to 1.0] — The median was not estimated due to low number of participants (as there were less than 3 participants).

9. Secondary Outcome: Time to Onset of Symptom Relief With Faces Pain Scale-Revised (FPS-R) Scores for Participants of 4 Years Age and Older
Description: The time to onset of symptom relief, defined as the duration of time in hours from the time of icatibant administration to the earliest time at which the post-treatment score improved by at least 1 level. Participants of 4 years age and older self-assessed their HAE-related pain using the FPS-R instrument. FPS-R is a self-reported measure used to assess the intensity of children's pain and it is scored using a 0 to 10 scale (0=no pain to 10=very much pain).
Time Frame: Baseline, and post dose on Day 1
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: hours
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
hours | NA [0.9 to 1.0] — The median was not estimated due to low number of participants (as there were less than 3 participants).

10. Secondary Outcome: Time to Onset of Symptom Relief by Faces, Legs, Activity, Cry, and Consolability (FLACC) Scale Assessed by Investigator for Participants of Younger Than 4 Years Age
Description: The time to onset of symptom relief, defined as the earliest time at which a 20% improvement is observed in the total post-treatment score. Participants of younger than 4 years age underwent investigator assessment of HAE-related pain (cutaneous, abdominal, and laryngeal) using the FLACC compartmental pain scale. Each of the 5 categories were scored from 0 to 2. Face(F): 0 (no particular expression/smile) - 2 (frequent to constant frown clenched jaw quivering chin); Legs(L): 0 (normal position/relaxed) - 2 (kicking/legs drawn up); Activity(A): 0 (lying quietly, normal position, moves easily) - 2 (arched rigid/jerking); Cry(C): 0 (No cry [awake/asleep]) - 2 (crying steadily/screams/sobs or frequent complaints); Consolability(C): 0 (content/relaxed) - 2 (difficult to console/comfort), resulting in a total score between 0 and 10.
Time Frame: Baseline, and post dose on Day 1
Population: As there were no participants between 2 to <4 years of age enrolled in this study, data was not collected for this outcome measure.
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Participants Who Were Treated With Rescue Medication During Study
Description: Rescue medication included therapies for HAE used for HAE attack and symptomatic treatment used in order to improve symptoms of angioedema (eg, pain and nausea).
Time Frame: Up to approximately 6 months
Population: Safety analysis set was defined as all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
Participants | 0

12. Secondary Outcome: Number of Participants With Worsened Intensity of Clinical HAE Symptoms Between 2 and 4 Hours After Treatment With SC Icatibant Using Investigator-Rated Symptom Scores
Description: Investigator-rated symptom score was used for assessment and scoring of cutaneous, abdominal, and laryngeal symptoms of acute HAE attacks related to daily activities. The score ranged from 0 to 4 and each number of scores means following; 0 = none; absence of symptoms, 1 = mild (no to mild interference with daily activities), 2 = moderate (moderate interference with daily activities), 3 = severe (severe interference with daily activities), 4 = very severe (very severe interference with daily activities).
Time Frame: From 2 hours post-dose to 4 hours post-dose
Population: Full analysis set was defined as all participants who had received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
Participants | 0

13. Secondary Outcome: Time to Initial Symptom Improvement Reported by Investigator
Description: Time to initial symptom improvement reported by investigator, was defined as the duration of time in hours from icatibant administration until the time when overall participant improvement was first noted by investigator.
Time Frame: Up to 8 hours post dose (or till the onset of HAE attacks were resolved)
Population: Full analysis set was defined as all participants who had received at least 1 dose of study drug.
Measure: Median (Full Range); unit: hours
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
hours | NA [0.3 to 1.0] — The median was not estimated due to low number of participants (as there were less than 3 participants).

14. Secondary Outcome: Time to Initial Symptom Improvement Reported by Participant
Description: Time to initial symptom improvement reported by participant, defined as the duration of time in hours from icatibant administration until the time when overall participant improvement was first noted by participant, participant's parent or participant's legal guardian.
Time Frame: Up to 8 hours post dose (or till the onset of HAE attacks were resolved)
Population: Full analysis set was defined as all participants who had received at least 1 dose of study drug.
Measure: Median (Full Range); unit: hours
Groups:
- TAK-667 10-30 mg: TAK-667 five-weight-band dosing of up to maximum of 30 mg injection, subcutaneously SC, once on Day 1, and if necessary (there was insufficient relief or worsening of symptoms), up to two additional doses with a time interval of at least 6 hours between doses within 48 hours of initial injection per attack for up to 3 HAE attacks till the end of study (approximately 6 months). The dose of TAK-667 depended upon the participant's body weight (10 mg for 12 kg to 25 kg, 15 mg for 26 kg to 40 kg, 20 mg for 41 kg to 50kg, 25 mg for 51 kg to 65 kg, 30 mg for >65 kg).
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
hours | NA [0.3 to 1.0] — The median was not estimated due to low number of participants (as there were less than 3 participants).

15. Secondary Outcome: Plasma Concentration for TAK-667
Time Frame: Day 1 pre-dose and at multiple timepoints post-dose
Population: Safety analysis set was defined as all participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: ug/l
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
ug/l
  Baseline (pre-dose) | 0 [0 to 0]
  0.5 hours postdose | NA [962 to 978] — The median was not estimated due to low number of participants (as there were less than 3 participants).
  1 hour postdose | NA [856 to 882] — The median was not estimated due to low number of participants (as there were less than 3 participants).
  2 hours postdose | NA [401 to 410] — The median was not estimated due to low number of participants (as there were less than 3 participants).
  4 hours postdose | NA [38.8 to 68.9] — The median was not estimated due to low number of participants (as there were less than 3 participants).

16. Secondary Outcome: Plasma Concentration for TAK-667 Metabolite M-I
Time Frame: Day 1 pre-dose and at multiple timepoints post-dose
Population: Safety analysis set was defined as all participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: ug/l
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
ug/l
  Baseline (pre-dose) | 0 [0 to 0]
  0.5 hours postdose | NA [103 to 106] — The median was not estimated due to low number of participants (as there were less than 3 participants).
  1 hour postdose | NA [187 to 223] — The median was not estimated due to low number of participants (as there were less than 3 participants).
  2 hours postdose | NA [220 to 247] — The median was not estimated due to low number of participants (as there were less than 3 participants).
  4 hours postdose | NA [124 to 137] — The median was not estimated due to low number of participants (as there were less than 3 participants).

17. Secondary Outcome: Plasma Concentration for TAK-667 Metabolite M-II
Time Frame: Day 1 pre-dose and at multiple timepoints post-dose
Population: Safety analysis set was defined as all participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: ug/l
Arm/Group | TAK-667 10-30 mg
Number analyzed (Participants) | 2
ug/l
  Baseline (pre-dose) | 0 [0 to 0]
  0.5 hours postdose | NA [103 to 116] — The median was not estimated due to low number of participants (as there were less than 3 participants).
  1 hour postdose | NA [184 to 216] — The median was not estimated due to low number of participants (as there were less than 3 participants).
  2 hours postdose | NA [227 to 276] — The median was not estimated due to low number of participants (as there were less than 3 participants).
  4 hours postdose | NA [147 to 151] — The median was not estimated due to low number of participants (as there were less than 3 participants).

ADVERSE EVENTS:
Time Frame: Up to approximately 6 months
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Data for injection site reactions were collected separately from general reports of AEs. As pre-defined in the protocol, an injection site reaction not meeting SAE criteria was not required to be reported additionally as an AE.
Arm/Group | TAK-667 10-30 mg
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Due to the low number of participants enrolled, the efficacy and pharmacokinetic data were not summarized to avoid risk of identification of the participant, only safety data was summarized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT04654351/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/51/NCT04654351/SAP_001.pdf